CLINICAL TRIAL: NCT03102411
Title: Impact of Diet on Functional Gastrointestinal Symptoms; a National Population Based Survey
Brief Title: Impact of Diet on Functional Gastrointestinal Symptoms
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-006
Record Dates: First submitted 2017-03-14; First posted 2017-04-05 (Actual); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-05

CONDITIONS: Gastrointestinal Disorder, Functional
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional survey study is to determine the prevalence of functional gastrointestinal (GI) disorders in the general population and to describe common triggers for food-related GI symptoms.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders, involving symptoms such as gas/bloating, diarrhea, constipation and abdominal pain, are estimated to impact between 35 and 45 million Americans, an overwhelming 15-20% of the population. These symptoms are responsible for upwards of 20 billion dollars in healthcare costs and extensive loss of quality of life for sufferers. Moreover, many patients suffer in silence, with 67% of subjects waiting more than a year before treatment, and 11% waiting over 10 years. Irritable bowel syndrome is the most prevalent functional gastrointestinal disorder, and several recent studies support the idea that dietary modifications may be key to alleviating this condition.

The purpose of this study is to document gastrointestinal symptoms among the US population, as well as to ascertain awareness and utilization of dietary treatments that exist.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Visual impairment
* Inability to read
* Inability to understand English
* Inability to use a computer to respond to questions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General popultion in the United States
Sampling Method: Non-Probability Sample
Enrollment: 1881 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The online survey took place from 3/9/2017 to 3/11/2017 through SurveyMonkey® (Palo Alto, CA, USA). The survey was distributed securely to a representative sample of the US population. 1881 subjects responded to the survey with 1718 completing all the questions (91% completers).
Groups:
- GI Symptoms Survey: The survey participants are men and women between the ages of 18 and 80 in the United States
Period: Overall Study
Arm/Group | GI Symptoms Survey
Started | 1881
Completed | 1718
Not Completed | 163

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: Out of 1881 subjects, 163 didn't completed the survey questionnaire and excluded from the data provided by SurveyMonkey. Descriptive statistics and data analysis were performed based on the data of 1718 subjects.
Groups:
- GI Symptoms Survey Population: The Survey participants are men and women between the ages of 18 and 80 in the United States
Arm/Group | GI Symptoms Survey Population
Number analyzed (Participants) | 1718
Age, Customized [Count of Participants; unit: Participants]
  18-30 years | 347
  31-45 years | 506
  46-60 years | 502
  61-80 years | 351
  Prefer not to answer | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 8 subject didn't answer the question of asking "Gender".
  Participants
    number analyzed (Participants) | 1710
    Female | 911
    Male | 799
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 1365
  African American/Black | 111
  Native American | 21
  Hawaiian or Pacific Islander | 10
  Asian | 70
  Prefer not to answer | 41
  Other | 100
Region of Enrollment [Number; unit: participants]
  United States | 1718

OUTCOME MEASURES:

1. Primary Outcome: Most Common Triggers for Food-related GI Symptoms (Top 5)
Description: Percentages for foods chosen as triggers ( a subject can check more than one answer - Bread, Oats, Chili, Corn, Onion, Garlic, Beans, Chocolate, Fried or greasy foods, Eggs, Soy, Red meat, Fish or shellfish, Dairy products, Nuts and seeds, Apples, Bananas, Citrus fruit, Alcohol, Coffee, Carbonated drinks, Sugar-free gum)
Time Frame: During the past 3 months before the survey
Measure: Count of Participants; unit: Participants
Groups:
- GI Symptom Survey Population: The survey participants are men and women between the ages of 18 and 80 in the United States.
Arm/Group | GI Symptom Survey Population
Number analyzed (Participants) | 1718
Participants
  Fried or greasy foods | 881
  Dairy products | 494
  Beans | 469
  Chili peppers | 460
  Alcohol | 354

2. Secondary Outcome: Self-reported Functional GI Disorders
Description: Percentages of self-reported functional GI disorders ( a subject can check more than one answer - Acid reflux (GERD), Irritable bowel syndrome (IBS), Celiac disease, Inflammatory bowel disease - Crohn's or Ulcerative Colitis, Diverticulities, Gastroparesis, Leaky gut, small intestinal bacterial overgrowth (SIBO), None of the above)
Time Frame: During the past 3 months before the survey
Measure: Count of Participants; unit: Participants
Arm/Group | GI Symptoms Survey
Number analyzed (Participants) | 1718
Participants
  Acid reflux (GERD) | 411
  Irritable bowel syndrome (IBS) | 161
  Celiac diseas | 23
  Inflammatory bowel disease | 33
  Diverticulitis | 72
  Gastroparesis | 26
  Leaky gut | 20
  Small intestinal bacterial overgrowth (SIBO) | 12
  None of the above | 1116

ADVERSE EVENTS:
Description: This is a survey study and collecting adverse event data is not applicable to this study.
Arm/Group | GI Symptoms Survey Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03102411/Prot_SAP_000.pdf